CLINICAL TRIAL: NCT00619762
Title: A Multicenter, Prospective, Open-Label Study to Assess the Clinical Outcomes of LTM Use in Two-Stage Breast Reconstruction Immediately Post Mastectomy
Brief Title: Immediate Postmastectomy Breast Reconstruction (Strattice Breast)
Status: Completed | Type: Observational
Sponsor: LifeCell (Industry)
Responsible Party: Sponsor
Other Study IDs: LFC2007.01.01
Record Dates: First submitted 2008-01-11; First posted 2008-02-21 (Estimated); Results first posted 2013-05-15 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-10

CONDITIONS: Breast Cancer
Keywords: Breast reconstruction
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tissue sample
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: LTM - a porcine-based surgical mesh — Use of LTM to support weak and/or absent soft tissue to facilitate immediate breast reconstruction postmastectomy

SUMMARY:
This prospective, multicenter, open-label study will assess the clinical outcomes of the LTM product in three planned analyses. The primary objective of this study is to prospectively assess the clinical outcomes associated with the use of LTM in two-stage (expander then permanent implant) immediate post-mastectomy breast reconstruction.

DETAILED DESCRIPTION:
nothing to add

ELIGIBILITY:
Inclusion Criteria:

* A candidate for immediate, two-stage breast reconstruction using LTM following a skin sparing mastectomy
* An ASA Physical Status Classification5 of 1 or 2 (see App I)
* Estimated life expectancy > 1 year

Exclusion Criteria:

* Clinically significant systemic disease
* Received inductive chemo-therapy within 2 months prior to mastectomy or radiation therapy to the region at any time
* Predicted excised breast mass of >750 gms
* Co-morbid factors which predispose to postoperative infection, such as insulin dependent diabetes, smoking, chronic steroid use, malnourishment, or co-existent infection
* Need for tissue flap in addition to expander
* History of alcohol abuse, illicit drug use, significant mental illness, physical dependence to any opioid, or drug abuse or addiction
* Enrollment or plans to enroll in another clinical trial during this study that would affect the patient's safety or results of this trial
* Any of the conditions identified within the labeled contraindications, i.e. sensitivity to porcine derived products or polysorbate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women undergoing two-stage immediate breast reconstruction following a skin sparing mastectomy will be recruited from up to ten (10) participating centers
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2007-10; Primary Completion 2009-10 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Franz, MD, Study Director — LifeCell
Locations (5):
- United States (5):
  - Washington D.C., District of Columbia
  - Chicago, Illinois
  - Great Neck, New York
  - Willow Grove, Pennsylvania
  - McLean, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 17 women were identified & consented to participate in the study. All were enrolled and received study product. Of the 17 women, 5 underwent unilateral reconstruction and 12 underwent bilateral reconstruction for a total of 29 breasts evaluated in the study. Patients were recruited from Hospital settings in PA, IL, Washington DC, NY, and VA.
Pre-assignment Details: This study was a prospective, multicenter, open-label study with no control arm. All enrolled women/breasts remained in the study through expander/implant exchange up through the Month 3 post-exchange visit.
Groups:
- LTM - Porcine Acellular Dermal Matrix in Breast Reconstruct: This was a single arm sudy without a control arm
  Use of LTM to reinforce weak tissue in two-stage (expander then permanent implant) immediate post-mastectomy breast reconstruction.
Period: Overall Study
Arm/Group | LTM - Porcine Acellular Dermal Matrix in Breast Reconstruct
Started | 17 ((29 breasts) First patient implanted 10/23/2007)
Completed | 14 ((25 breasts) last patient visit 11/09/2009)
Not Completed | 3

BASELINE CHARACTERISTICS:
Groups:
- LTN - Porcine Acellulare Dermal Matrix in Breast Recon: This was a single arm sudy without a control arm LTM used to reinforce weak tissue in breast reconstruction surgery
Arm/Group | LTN - Porcine Acellulare Dermal Matrix in Breast Recon
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Secondary Outcome: Severity of Local Inflammation at and Around the Surgical Site
Description: The Inflammatory response was evaluated by each of the four cardinal signs: erythema, edema, pain and heat, using standard scales for the evaluation of each sign and inflammation as a whole was assessed using a model (AIR Score) which took into account the scores assigned to each of the four signs. A mean score is provided at each timepoint.The minimum total possible score is 4 (less inflamation) and the maximum total possible score is 8 (more inflammation).
Time Frame: Postoperative Day 7, 14, 21, 30 days
Population: Total breasts enrolled were 29. Day 7, N = 28 breasts available Day 14, N = 27 breasts available Day 21, N = 27 breasts available Day 30, N = 25 breasts available
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Breasts
Groups:
- Treatment Arm: all available patients/breasts who completed specified visit
Arm/Group | Treatment Arm
Number analyzed (Participants) | 17
Number analyzed (Breasts) | 29
units on a scale
  Day 7 (n=28) Final AIR Score | 5.71 (1.11)
  Day 14 (n=27) Final AIR Score | 5.55 (1.28)
  Day 21 (n=27) Final AIR Score | 5.07 (1.47)
  Day 30 (n=25) Final AIR Score | 4.84 (1.10)

2. Primary Outcome: Histology Sample Evaluations Assessing Incorporation of StratticeTM Reconstructive Tissue Matrix
Description: Evaluation of 3 histology parameters, fibroblast infiltration, immune cell response & revascularization, expressed as frequency distributions. Samples evaluated for presence of fibroblasts (cellularity), neovascularization & immune cell response using 4 pt scale. Fibroblast Infiltration: 1=None,2=Few,sparse,3=Moderate,4=Dense. Revascularization:1=None,2=Few randomly dispersed capillaries,3=Moderate; mostly homogenous distribution of new vessels,4=Significant,uniformly distributed vessels; both capillaries and arterioles. Immune Cell response: 1= None,2=Few,normal healing response,3=Moderate,4=Significant;above expected presence for healing. 4 high power(HP)fields reviewed & if uniform in appearance/cellular distribution, 4 considered representative of sample as a whole. If non-uniform distribution observed, 3 HP fields of "sparse or light" distribution & 3 HP fields of dense distribution counted & results averaged. Tissue sample then assessed for overall acellularity & expressed as %.
Time Frame: At the time of expander/implant exchange (Stage II),
Population: All implanted patients enrolled in the study were included in the analysis
Measure: Number; unit: percentage of breasts
Units Other Than Participants: Breasts
Groups:
- Treatment Arm: All implanted patients in the study, that is 29 breasts in 17 patients
Arm/Group | Treatment Arm
Number analyzed (Participants) | 17
Number analyzed (Breasts) | 29
percentage of breasts
  Fibroblast Infiltration Percent = None | 0
  Fibroblast Infiltration Percent = Few | 82.8
  Fibroblast Infiltration Percent = Moderate | 17.2
  Fibroblast Infiltration Percent=Significant (dense | 0
  Immune Cell Response Percent = None | 3.4
  Immune Cell Response Percent = Few | 13.7
  Immune Cell Response Percent = Moderate | 10.3
  Immune Cell Response Percent = Significant | 72.4
  Revascularization Percent = None | 65.5
  Revascularization Percent = Few | 31
  Revascularization Percent = Moderate | 3.4
  Revascularization Percent = Significant | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from day of implantation through the 12 month visit
Arm/Group | Treatment Arm
Serious Adverse Events (participants affected / at risk) | 3/17
Other Adverse Events (participants affected / at risk) | 2/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=17)
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) — On POD 7, Mediport was placed. During placement, a pneumothorax occurred. A chest tube was placed to reinflate lung and was removed 5 days later. Event was not considered related to device & resolved without sequelae on POD 12.
Infection (Infections and infestations) | 1 (1) — On POD 21, erythema of lower breast flap was noted & antibiotics initiated. After 2 wk course of antibiotics, erythema had resolved & antibiotics discontinued. Event was considered possibly related to device & resolved without sequelae on POD 36.
post operative bleeding (Vascular disorders) | 1 (1) — After breast reconstruction, severe bleeding was noted while in recovery rm. Subject returned to OR for control of bleeding by ligation of small artery. Event was not considered to be related to device & resolved without sequelae on day of surgery.
Breast deformity (Skin and subcutaneous tissue disorders) | 1 (1) — On POD 229, subject noted to have significant deformity of breast/lack of subcutaneous tissue.Subject received fat grafting.Event was not considered related to device & subject recovered without sequelae.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=29)
infection (Infections and infestations) | 2 (2) — Infection of breast flap on POD 53 that was possibly related to device and resolved without sequelae Infection of breast flap on POD 37 that ws possibly Resolved to device and resolved without sequelae

LIMITATIONS AND CAVEATS:
Small number of subjects and breasts analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No